CLINICAL TRIAL: NCT00437255
Title: An Evaluation of the Efficacy, Safety, Preference and Duration of Response of Clobex® (Clobetasol Propionate) Spray and Taclonex® (Calcipotriene 0.05%/Betamethasone Dipropionate 0.064%) Ointment in Subjects With Stable Plaque Psoriasis
Brief Title: Efficacy, Safety, Preference and Response Duration of Clobex® Spray and Taclonex® Ointment in Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma Laboratories, L.P.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10034
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-04

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Clobetasol; calcipotriene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Clobex® Spray
  Interventions: Drug: Clobetasol Propionate, 0.05%
- 2 (Active Comparator): Taclonex® Ointment
  Interventions: Drug: Calcipotriene and betamethasone dipropionate ointment

INTERVENTIONS:
Drug: Clobetasol Propionate, 0.05% — Topical, twice daily for 4 weeks
  Other Names: Clobex® Spray
  Arms: 1
Drug: Calcipotriene and betamethasone dipropionate ointment — Topical, once daily
  Other Names: Taclonex® Ointment
  Arms: 2

SUMMARY:
Evaluate the efficacy of Clobex® Spray as compared to Taclonex® Ointment in terms of Overall Disease Severity and Investigator Global Assessment.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe psoriasis involving 3-20% of the body surface area

Exclusion Criteria:

* Subjects who have surface area involvement too large that would require more than 50 grams per week of Clobex® Spray or more than 100 grams per week of Taclonex® Ointment
* Subjects having psoriasis that involves the scalp, face, or groin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Overall Disease Severity | End of treatment (Week 4)
Tolerability assessments, incidence of adverse events | Baseline, Weeks 1, 2, 4 and 8

SECONDARY OUTCOMES:
Overall Disease Severity | Weeks 1, 2 and 8
Investigator Global Assessment | End of treatment (week 4) and Weeks 1, 2 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma Laboratories, LP
Locations (4):
- United States (4):
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., Bryan, Texas
  - Baylor Research Institute, Dallas, Texas